CLINICAL TRIAL: NCT04543331
Title: OBservationaL stUdy to Evaluate Fluid reSolution and Effectiveness in Patients Receiving Beovu (Brolucizumab) Under KeY Treatment Schemes in Neovascular Age-related Macular Degeneration and Visual Impairment Due to Diabetic Macular Edema
Brief Title: Observational Study to Evaluate Fluid Resolution and Effectiveness in Patients Receiving Beovu in Neovascular Age-related Macular Degeneration and Visual Impairment Due to Diabetic Macular Edema
Acronym: BLUE SKY
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258ADE02
Record Dates: First submitted 2020-09-04; First posted 2020-09-10 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Neovascular Age-related Macular Degeneration (nAMD); Diabetic Macular Edema (DME)
Keywords: Beovu; Brolucizumab; nAMD; DME; non-interventional trial; effectiveness; fluid resolution; treatment intervals; real world study
MeSH Terms: interventions — brolucizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- treatment naïve patients: Patients being the first time treated for nAMD or DME
  Interventions: Drug: brolucizumab
- pre-treated patients: Patients already being treated for nAMD or DME
  Interventions: Drug: brolucizumab

INTERVENTIONS:
Drug: brolucizumab — There is no treatment allocation. Patients administered Brolucizumab by prescription that have started before inclusion of the patient into the study will be enrolled.

SUMMARY:
This study is a prospective, non-interventional, multicenter, open-label study in nAMD and DME patients being treated with brolucizumab according to the EU SmPC.

An observational study design, without a strict, mandated visit schedule or mandated treatment regimen was chosen as the most appropriate to collect available data in a real life setting. For that reason, this NIS does not impose a therapy protocol, diagnostic/therapeutic procedure or a visit schedule. The diagnostic or monitoring procedures are only those ordinarily applied to the therapeutic strategy and to routine clinical care and will take place as per investigator's discretion. This includes e.g. visit frequency, injection frequency and types of assessments performed - only data from routine medical practice will be collected as part of the study.

DETAILED DESCRIPTION:
BLUE SKY consists of the nAMD-related module BIRL (Brolucizumab In Real Life) and two general, indication-related study modules "BLUE SKY AMD" and "BLUE SKY DME".

Patients will be enrolled at approximately 55 centers, which will be representatively distributed amongst the 16 German federal states. This will ensure to reflect all state-specific health insurance laws and guidelines. Naïve and pre-treated patients will be included after decision to start treatment with brolucizumab and consent is given.

All patients will be documented either in the AMD or DME-module (Full Analysis Set).

For the BIRL module, only naïve nAMD patients enrolled in approximately 7 selected centers will be documented. All these centers are equipped with the Zeiss PlexElite OCT-A, needed to assess and analyze BIRL specific objectives in a comparable setting. Only images from routine medical practice will be collected as part of the study. The study eye will be defined as the first eye treated during the study, the other eye will be considered as fellow eye.

If both eyes are treated at baseline, the eye with the worse VA will be chosen as the study eye (if VA is measured equal, the treating ophthalmologist defines the study eye upon his discretion).

The prospective observation period per patient will be up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

The unit of analysis is patient-eye, i.e. all criteria should be applied to the study eye, unless otherwise specified. Patients will be included in the study if they fulfil the following requisites:

1. Diagnosis of nAMD or visual impairment due to DME
2. Male and Female nAMD and DME patients with ≥18 years of age at index
3. Decision to treat with brolucizumab at baseline visit
4. Signed written informed consent
5. Patients for whom a therapy with brolucizumab is medically indicated
6. Intraretinal and/or subretinal fluid affecting the central subfield of the study eye at Screening

Exclusion Criteria:

1. Patients that have any contraindication or are not eligible for treatment with brolucizumab as according to the SmPC
2. Patients treated for RVO or CNV other than nAMD
3. Receipt of any anti-VEGF treatment other than brolucizumab in the study eye at index date
4. Central subfield of the study eye affected by fibrosis or geographic atrophy or total area of fibrosis >50% of the total lesion (nAMD)
5. Any active intraocular or periocular infection or active intraocular inflammation in either eye at index date
6. Patients who have been on anti-VEGF treatment for longer than 3 years (before index date)
7. Any medical or psychological condition in the treating physician's opinion which may prevent the patient from the 24 months study participation
8. Patients participating in parallel in an interventional clinical trial
9. Patients participating in parallel in any other NIS generating primary data for an anti-VEGF drug
10. Laser photocoagulation (focal/grid or panretinal) in the study eye during the 3-month period prior to baseline
11. Prior use of intraocular or periocular corticosteroids in the study eye provided at least 4 months prior to baseline
12. Pregnancy and breast-feeding

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated for nAMD or DME with brolucizumab will be enrolled in the study upon signing an informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 572 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Percentage of patients' eyes that are absent of subretinal fluid (SRF) and intra-retinal fluid (IRF) | Month 12
  This outcome measure is part of the BLUE SKY AMD module. This primary study objective will be addressed considering treatment naïve and pre-treated patient eyes, analyzed as two independent groups (naïve and switch).
Mean change in visual actuity (VA) under clinic specific routine treatment schemes | Baseline, month 12
  This outcome measure is part of the BIRL module. This primary study objective will be addressed considering treatment naïve patient eyes.
  Index date (Baseline): defined as the date of the first anti-VEGF injection (brolucizumab) in patient eye.
Morphological CNV-Changes under clinic specific routine treatment schemes | Baseline, month 12
  This outcome measure is part of the BIRL module. This primary study objective will be addressed considering treatment naïve patient eyes.
  Index date (Baseline): defined as the date of the first anti-VEGF injection (brolucizumab) in patient eye.
Percent of patients maintained on q12w dosing after loading through Week 52 | After loading, month 12
  This outcome measure is part of the BLUE SKY DME module. This primary study objective will be addressed considering treatment naïve patient eyes included in the study.
Change in interval length from last interval before switch (baseline) to last interval at end of follow-up (12 months) | Baseline, month 12
  This outcome measure is part of the BLUE SKY DME module. This primary study objective will be addressed considering pre-treated patient eyes. Index date (Baseline): defined as the date of the first anti-VEGF injection (brolucizumab) in patient eyes.

SECONDARY OUTCOMES:
Characterize nAMD patients who initiated treatment with brolucizumab with the respect to baseline characteristics | Baseline
  nAMD patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Evaluate anatomical parameters during treatment with brolucizumab | Up to month 24
  nAMD patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan.
Evaluate VA change from baseline during treatment with brolucizumab | Baseline, month 24
  nAMD patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan.
Estimate number of anti-VEGF injections, visits and injection intervals | Up to month 24
  nAMD patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Estimate percentage of switchers during first 6 months and characterize switchers | Baseline, month 6
  nAMD patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Estimate discontinuation rate and time to discontinuation | Month 1-12 and 13-24
  nAMD patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Assess retreatment criteria | Up to month 24
  nAMD patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Estimate the number of OCT | Month 1-12 and 13-24
  nAMD patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Assess the safety of brolucizumab | Up to month 24
  nAMD patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Evaluate anatomical effectiveness | Up to month 24
  naive nAMD patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Evaluate treatment intervals | Up to month 24
  naive nAMD patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Describe implementation of treatment schemes into clinical practice | Up to month 24
  naive nAMD patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Evaluate morphological changes under brolucizumab treatment using multimodal imaging | Up to month 24
  naive nAMD patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Percentage of patient's eyes with absence of IRF and/or SRF at month 12 (naive and switch) | Month 12
  DME patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Evaluate anatomical parameters during treatment with brolucizumab | Month 1-12 and 13-24
  DME patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Characterize VA change from baseline during treatment with brolucizumab | Month 1-12 and 13-24
  DME patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Estimate discontinuation rate during first year of brolucizumab treatment | Baseline, month 12
  DME patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Estimate time to discontinuation (persistence) | Up to month 24
  DME patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Estimate the treatment burden | Month 1-12 and 13-24
  DME patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Estimate the number of OCT and the number of visits with/without OCT | Month 1-12 and 13-24
  DME patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan.
Assess safety of brolucizumab | Up to month 24
  DME patients. Detailed Outcome Measure will be defined in the Statistical Analysis Plan.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (38):
- Germany (38):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Osnabrück, Lower Saxony
  - Novartis Investigative Site, Rostock, Mecklenburg-Vorpommern
  - Novartis Investigative Site, Trier, Rhineland-Palatinate
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Schneeberg, Saxony
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Aschersleben
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Breisach
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Esslingen am Neckar
  - Novartis Investigative Site, Glauchau
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Hösbach
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Marienberg
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neubrandenburg
  - Novartis Investigative Site, Neuburg am Inn
  - Novartis Investigative Site, Saarbrücken
  - Novartis Investigative Site, Schönebeck
  - Novartis Investigative Site, Stralsund
  - Novartis Investigative Site, Sulzbach
  - Novartis Investigative Site, Torgau
  - Novartis Investigative Site, Waren
  - Novartis Investigative Site, Würzburg

IPD SHARING:
Plan to Share IPD: No